CLINICAL TRIAL: NCT03026881
Title: An Open, Non-randomised, Multi-centre Phase I Study to Assess the Safety and Efficacy of Fluzoparib Given in Combination With Apatinib and Paclitaxel in the 2nd Line Treatment of Patients With Recurrent or Metastatic Gastric Cancer
Brief Title: A Study of Fluzoparib Given in Combination With Apatinib and Paclitaxel in Gastric Cancer Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FZPL-I-103-GC
Record Dates: First submitted 2016-12-21; First posted 2017-01-20 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Recurrent and Metastatic Gastric Cancer
Keywords: PARP inhibitor; VEGFR inhibitor; Combination therapy; Gastric cancer
MeSH Terms: conditions — Recurrence; Stomach Neoplasms | interventions — fluzoparib; apatinib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluzoparib + Apatinib + Paclitaxel (Experimental)
  Interventions: Drug: Fluzoparib; Drug: Apatinib; Drug: Paclitaxel

INTERVENTIONS:
Drug: Fluzoparib — Fluzoparib either at 20,30,40mg twice daily,capsule oral.
  Other Names: SHR3162
Drug: Apatinib — Oral
Drug: Paclitaxel — Intravenous injection

SUMMARY:
Fluzoparib is an oral potent, selective PARP-1 and PARP-2 inhibitor; Apatinib is an oral selective VEGFR inhibitor. This open-label, dose finding phase I trial studies the tolerability and the best dose of Fluzoparib in combination with apatinib and paclitaxel and to see how well this three drugs work together in the treatment of patients with recurrent and metastatic gastric cancer who progress following first-line therapy. The safety and efficacy of fluzoparib in combination with apatinib and paclitaxel will be explored.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status of 0 to 1.
* Life expectancy of more than 12 weeks.
* Histologically or cytologically confirmed gastric adenocarcinoma( adenocarcinoma of the gastroesophageal junction included).
* Recurrent or metastatic gastric cancer that has progressed following first line-therapy.
* At least one lesion (measurable and/or non-measurable) that can be accurately assessed by imaging (CT/MRI) at baseline
* Subjects who have overall good overall general condition.
* Signed informed consent.

Exclusion Criteria:

* Subjects who received any previous treatment with any PARP inhibitors.
* Subjects who received any previous treatment with any taxanes.
* More than one prior chemotherapy regimen for the treatment of gastric cancer in the metastatic or recurrent setting.
* Less than 4 weeks from the last clinical trial.
* Less than 2 weeks from the last radiotherapy, chemotherapy, surgery, hormone treatment and target therapy.
* Unstable hypertension.
* Subjects that are unable to swallow, or dysfunction of gastrointestinal absorption.
* Subjects with brain metastases.
* Subjects with uncontrolled hypokalemia and hypomagnesemia before study entry.
* Subjects with a known hypersensitivity to fluzoparib, apatinib, paclitaxel or any of the excipients of the product.
* Ongoing infection (determined by investigator).
* History of immunodeficiency, including HIV-positive, suffering from other acquired, congenital immunodeficiency disease, or history of organ transplantation.
* Subjects who can not interrupt the using of the drugs that may cause QT prolongation during study.
* Pregnant or breast-feeding women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-04 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
DLT and safety: Adverse Events (AEs), physical examination, vital signs including blood pressure (BP), pulse, electrocardiogram (ECG) and laboratory findings including clinical chemistry, hematology, urinalysis. | through study completion, an average of 6 months
  DLT and safety defined by CTC version 4.0

SECONDARY OUTCOMES:
Best of ORR | through study completion, an average of 6 months
Overall Response Rate (ORR) | through study completion, an average of 6 months
Disease Control Rate (DOR) | through study completion, an average of 6 months
Time to Progression (TTP) | From date of enrollment until the date of first objective progression, assessed up to 9 months
Progression Free Survival (PFS) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, an average of 6 months
Maximum plasma concentration (Cmax) | Up to 33 days
Terminal half life (t1/2) | Up to 33 days
Area under the plasma concentration-time curve (AUC） | Up to 33 days
Volume of distribution (V/F) | Up to 33 days
Plasma Clearance (CL/F) | Up to 33 days

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Military Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided